CLINICAL TRIAL: NCT04928911
Title: Expectations About the COVID-19 Vaccines
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AUvac
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Vaccine Adverse Reaction
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults receiving COVID-19 vaccine: Adults about to receive a COVID-19 vaccine fill out a questionnaire of potential predictors of side effect occurrence
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — Adults about to receive a COVID-19 vaccine fill out a questionnaire of potential predictors of side effect occurrence

SUMMARY:
This study collects information on expectations and attitudes towards the COVID-19 vaccines in participants about to receive a COVID-19 vaccine. This information will be linked to data on side effect occurrence collected in an independent study.

DETAILED DESCRIPTION:
General hypothesis: Negative expectations and attitudes towards the vaccine are associated with a higher risk of side effects

ELIGIBILITY:
Inclusion Criteria:

* Must have signed up to receive a COVID-19 vaccine in Denmark
* Participants are also a part of the ENFORCE study from which outcome data is obtained
* Must be able to read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults signed up to receive a COVID-19 vaccine in Denmark, who are also participating in the ENFORCE study
Sampling Method: Non-Probability Sample
Enrollment: 1176 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of local and systemic reactions (self-report) | 7 days after vaccination
  Data obtained from independent study
Rate of local and systemic reactions (self-report) | 14 days after vaccination
  Data obtained from independent study

SECONDARY OUTCOMES:
Grade 1-4 and serious adverse events | 3-6 months after vaccination
  Data obtained from independent study

CONTACTS AND LOCATIONS:
Overall Officials: Lene Vase, Study Chair — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No